CLINICAL TRIAL: NCT00836641
Title: Prospective Randomized Controlled Phase 4 Study on the Safety and Immunogenicity of Sequential Pneumococcal Immunization in Preschool Asthmatics
Brief Title: Safety and Immunogenicity of Sequential Pneumococcal Immunization in Preschool Asthmatics
Acronym: PAPSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Markus Rose, Professor of Paediatrics, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAPSI.FFM.3217
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
Keywords: preschool asthma; sequential pneumococcal immunization; immunogenicity; safety
MeSH Terms: conditions — Asthma | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pneumococcal immunization (2 mo) (Active Comparator): one dose of pneumococcal conjugate vaccine (prevenar) followed after 2 months by one dose of pneumococcal polysaccharide vaccine (pneumovax)
  Interventions: Biological: prevenar; Biological: pneumovax
- pneumococcal immunization (10 mo) (Active Comparator): one dose of pneumococcal conjugate vaccine (prevenar) followed after 10 months by one dose of pneumococcal polysaccharide vaccine (pneumovax)
  Interventions: Biological: prevenar; Biological: pneumovax

INTERVENTIONS:
Biological: prevenar — 7-valent pneumococcal conjugate vaccine
  Other Names: Prevnar, PCV-7
Biological: pneumovax — 23 valent pneumococcal polysaccharide vaccine
  Other Names: pneumopur, PPV-23

SUMMARY:
Asthma is a major health problem in preschool children. Infections by pneumococci a the most frequent cause of airway infections, which tend to cause worsening of asthma. Vaccination against pneumococci is recommended by scientific boards and the medical community, in order to reduce the burden of disease. Data on the immunogenicity and safety of pneumococcal immunization in preschool asthmatics are scarce.

DETAILED DESCRIPTION:
Respiratory infections are major triggers of exacerbations in preschool asthma. Many countries' guidelines recommend immunization against pneumococci for patients suffering from chronic airway disease. Also the interval between priming and booster is a matter of debate.

We immunize a large group of preschool asthmatics (2-5 years old) sequentially: one dose of seven-valent pneumococcal conjugate vaccine (PCV-7) followed by a single dose of 23-valent pneumococcal polysaccharide vaccine (PPV-23). We randomly assign half of the vaccinees to receive PPV-23 eight weeks after PCV-7 (group A), and the rest to a 10-month interval (group B). Pneumococcal antibody concentrations to serotype 4, 5, 6B, 7, 9V, 14, 18c, 19F, and 23F are determined initially, after two, and 12 months after PCV-7. Local and systemic reactions to each vaccine are recorded.

ELIGIBILITY:
Inclusion Criteria:

* asthma classified according to the Global Initiative on Asthma (GINA) °1-2

Exclusion Criteria:

* antecedent pneumococcal immunization

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, M.D., Principal Investigator — Goethe University Childrens Hospital

REFERENCES:
- [Background] Rose MA, Schubert R, Kujumdshiev S, Kitz R, Zielen S. Immunoglobulins and immunogenicity of pneumococcal vaccination in preschool asthma. Int J Clin Pract. 2006 Nov;60(11):1425-31. doi: 10.1111/j.1742-1241.2006.01093.x. PMID 17073839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11/2005-09/07: 70 outpatients (2-5-yo)with >3 asthma episodes during 12 months. Exclusion: pneumococcal immunization,severe/unstable asthma, systemic steroids, preterm birth (<37 weeks of gestation), low birthweight (<2500 g), major congenital abnormalities, and known intolerance towards ingredients of the pneumococcal vaccines.
Groups:
- Group A: Sequential Pneumococcal Immunzation (2 mo): one dose of pneumococcal conjugate vaccine followed after 2 months by one dose of pneumococcal polysaccharide vaccine
- Group B: Sequential Pneumococcal Immunization (10 mo): one dose of pneumococcal conjugate vaccine followed after 10 months by one dose of pneumococcal polysaccharide vaccine
Period: Overall Study
Arm/Group | Group A: Sequential Pneumococcal Immunzation (2 mo) | Group B: Sequential Pneumococcal Immunization (10 mo)
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A Pneumococcal Immunization (2 mo): one dose of pneumococcal conjugate vaccine followed after 2 months by one dose of pneumococcal polysaccharide vaccine
- Group B Pneumococcal Immunization (10 mo): one dose of pneumococcal conjugate vaccine followed after 10 months by one dose of pneumococcal polysaccharide vaccine
- Total: Total of all reporting groups
Arm/Group | Group A Pneumococcal Immunization (2 mo) | Group B Pneumococcal Immunization (10 mo) | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 34 | 70
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3 (0.5) | 3 (0.7) | 3 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  Germany | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of Pneumococcal Vaccination
Description: we performed pneumococcal serotype specific ELISA according to WHO's criteria for protective threshold values (>0.35 µg/ml).
Time Frame: 12 months
Population: we performed a power calculation in advance. To demonstrate a difference wit p<0.05, we would require 30 subjects per arm each. Thus and to allow potential drop-outs, we included 35 subjects per arm.
Measure: Geometric Mean (95% Confidence Interval); unit: [µg/ml]
Arm/Group | Group A Pneumococcal Immunization (2 mo) | Group B Pneumococcal Immunization (10 mo)
Number analyzed (Participants) | 36 | 34
[µg/ml] | 0.05 [0.01 to 5.00] | 0.05 [0.01 to 5.00]

2. Secondary Outcome: Number of Vaccinees With Adverse Events
Description: we evaluated the safety and tolerability of sequential pneumococcal immunization as to local and systemic adverse events.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Group A Pneumococcal Immunization (2 mo) | Group B Pneumococcal Immunization (10 mo)
Number analyzed (Participants) | 36 | 34
participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Overall Study Population: the whole study population was observed for adverse events.
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No